CLINICAL TRIAL: NCT02027727
Title: Individualized Infiximab Dosing-Proof of Concept Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Namita Singh, M.D., Attending Physician of Pediatrics IBD Center, Cedars Sinai Med Center, Cedars-Sinai Medical Center
Other Study IDs: Infiximab Dosing
Record Dates: First submitted 2013-12-09; First posted 2014-01-06 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: inflammatory bowel disease; infliximab; trough level; crohn's disease; ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No intervention: No intervention- this is an observational study of patients receiving Infliximab.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — no intervention- tihs is an observational study

SUMMARY:
The purpose of this study is to determine which early infliximab pharmacokinetic level is most associated with clinical remission at weeks 30 and 54 in pediatric IBD patients.

DETAILED DESCRIPTION:
Our aims are:

1. to determine which early pk level; week 6 (peak), week 8 (2 week) or week 14 (trough), is most associated with week 30 and 54 outcomes in pediatric IBD patients.
2. to determine if the forecasted PK determined by a newly developed Population PK Model software program is in agreement with the observed PK in IBD patients receiving infliximab.

Subject recruitment is limited to patients of the principal investigator only. Subjects will be approached for participation in the research in person during a routine clinic visit by a member of the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females on IFX
2. Patients with IBD
3. Age 6-23
4. Able to obtain consent

Exclusion Criteria:

1. Not receiving infliximab
2. On 10 mg/kg of IFX
3. Not able to obtain consent

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Males and females patients age 6 to 23
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-05 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Infliximab level and clinical remission at 54 weeks | 54 weeks
  Determine what level (peak, 2 week or trough) best correlates with clinical remission at week 54
  Clinical remission definition: PCDAI < 10 or CDAI < 150 for Crohn's disease, or partial Mayo <2 points and no sub-score > 1 for ulcerative colitis.
  Fischer exact testing will be done to determine what detectable IFX level (week 6, week 8 or week 14) is most associated with week 54 clinical remission.
  Wilcoxon rank sum test will be performed to determine the median level that is most associated with week 54 clinical remission.
  Regression tree analysis will be performed to determine the optimal infliximab level cut point that predicts week 54 clinical remission.
Infliximab level and clinical remission at 30 weeks | 30 weeks
  Determine what level (peak, 2 week or trough) best correlates with clinical remission at week 30
  Clinical remission definition: PCDAI < 10 or CDAI < 150 for Crohn's disease, or partial Mayo <2 points and no sub-score > 1 for ulcerative colitis.

SECONDARY OUTCOMES:
Agreement between pk profiles predicted by the PK model and actual (measured) pk profiles | 1 year
  Secondary outcomes
  1. Agreement between pk profiles predicted by the PK model and actual (measured) pk profiles for all patients with at least 6 months in between levels Analysis: Bland Altman test will be used to quantify the agreement between the two methods: Software pk model vs actual measured pk profiles
  2. Comparison of software selected dose regimens with actual dose regimens for cost and overall drug exposure (AUC and Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Namita Singh, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States